CLINICAL TRIAL: NCT07095075
Title: An Open-label Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LUCAR-DKS1 in Subjects With Relapsed/Refractory Autoimmune Diseases (r/r AID)
Brief Title: A Study of LUCAR-DKS1 in Subjects With Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LB2405-0001
Record Dates: First submitted 2025-06-23; First posted 2025-07-31 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: This study is a dose exploration study that employs an accelerated titration design combined with BF-BOIN, planned to investigate 5 dose groups. Dose Level1 （25×10^6 cells/kg) and Level 2(50×10^6 cells/kg)belong to the accelerated titration method for dose assessment, three dosage levels of 100×10^6 cells/kg, 200×10^6 cells/kg, and 400×10^6 cells/kg are assessed using the BOIN dose escalation and de-escalation rules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric antigen receptor NK cells (LUCAR-DKS1), single-dose for each subject. (Experimental): Experimental: chimeric antigen receptor NK cells (LUCAR-DKS1). Dose level1：25 millions /kg Dose level2：50 millions /kg Dose level3：100 millions /kg Dose level4：200 millions /kg Dose level5：400 millions /kg Totally 5 dose groups, each subject will be given a single-dose LUCAR-DKS1 cells infusion at a certain level, subject will be administered at day 1.
  Interventions: Biological: LUCAR-DKS1 NK cells

INTERVENTIONS:
Biological: LUCAR-DKS1 NK cells — Prior to the infusion of the LUCAR-DKS1 cells, subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine.

SUMMARY:
This is a prospective, single-arm, open-label and dose-escalation Investigator Initialed study to evaluate LUCAR-DKS1 in adult subjects with relapsed/refractory autoimmune diseases.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy profiles of LUCAR-DKS1, a chimeric antigen receptor (CAR) -NK cell therapy in subjects with relapsed/refractory autoimmune diseases. Patients who meet the eligibility criteria will receive LUCAR-DKS1 infusion. The study will include the following sequential stages: screening, pre-treatment (lymphodepleting chemotherapy), treatment LUCAR-DKS1 infusion) and follow-up.

ELIGIBILITY:
* Inclusion Criteria:

  1. Subjects voluntary agreement to provide written informed consent.
  2. Aged 18 to 70 years, either sex.
  3. Clinical laboratory values meet screening criteria.
  4. Positive test for CD19 and/ or BCMA

SLE:

* Meets at least 1 classification criteria≥6 months for SLE.
* At screening, antinuclear antibody, and/or anti-dsDNA antibody, and/or anti-Smith antibody should be positive.
* Fulfill relapsed/refractory SLE conditions.

AAV:

* Meets the 2022 ACR/EULAR classification criteria for AAV.
* Positive test for anti-MPO or p-ANCA or anti-PR3 or anti-MPO antibodies at screening.
* Fulfill relapsed/refractory AAV conditions.

SSc:

* Meets the 2013 ACR/EULAR classification criteria for SSc.
* At screening, mRSS is higher than 10.
* Fulfill relapsed/refractory SSc conditions.

IIM:

* Meets 2017 EULAR/ACR classification criteria for IIM.
* Positive test for myositis-associated antibodies or myositis-specific antibodies at screening.
* Fulfill relapsed/refractory IIM conditions. SjS：
* Meets the 2016 ACR/EULAR diagnostic criteria for SjS.
* Positive test for anti-SSA and/or anti-SSB antibodies at screening.
* Fulfill relapsed/refractory SjS conditions.

Exclusion Criteria:

1. Active infections such as hepatitis and tuberculosis.
2. Other autoimmune diseases.
3. Serious underlying diseases such as tumor, uncontrolled diabetes.
4. Female subjects who were pregnant, breastfeeding.
5. Those with a history of major organ transplantation.
6. Have received autologous cell therapy of any target before.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) . | About 2 years after LUCAR-DKS1infusion (Day 1)
  ≥Grade 1 clinical symptoms, laboratory test abnormalities, and clinical events that are possibly, likely, or definitely related to study treatment. Accessed by CTCAE5.0.
Incidence of dose-limiting toxicity (DLT) | About 2 years after LUCAR-DKS1 infusion (Day 1)
  DLTs are severe adverse events that refers to any untoward medical occurred in a subject participated in a clinical investigation, which have a causal relationship with the treatment and will limit the dose escalation.
Cmax | About 2 years after LUCAR-DKS1 infusion (Day 1)
  CAR positive NK cells in peripheral blood after LUCAR-DKS1 infusion, maximum concentration (Cmax).
Tmax | About 2 years after LUCAR-DKS1 infusion (Day 1)
  CAR positive NK cells levels in peripheral blood after LUCAR-DKS1 infusion, time to Cmax (Tmax).
AUC | About 2 years after LUCAR-DKS1 infusion (Day 1)
  CAR positive NK cells levels in peripheral blood after LUCAR-DKS1 infusion， area under the concentration-time curve (AUC) .
Recommended phase 2 dose regimen finding | About 2 years after LUCAR-DKS1 infusion (Day 1)
  Recommended phase 2 dose regimen established through dose exploratoration finding.

SECONDARY OUTCOMES:
SLE disease activity: Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | About 2 years after LUCAR-DKS1infusion (Day 1)
  Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) scores from baseline up to 2 years, a total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
SSc disease activity :Modified rodnan skin score(mRSS) | About 2 years after LUCAR-DKS1 infusion (Day 1)
  Change in modified Rodnan skin score (mRSS) from baseline up to 2 years in SSc patients. The mRSS is used to assess skin thickness and scope of SSc patients ,with a total score can fall between 0 and 51, with a higher score representing a more significant degree of skin involvement.
AAV disease activity： Birmingham vasculitis activity score (BVAS) | About 2 years after LUCAR-DKS1 infusion (Day 1)
  Change in Birmingham vasculitis activity score (BVAS) from baseline up to 2 years in patients with AAV. A total score can fall between 0 and 64, with a higher score representing a more significant degree of disease activity.
IIM disease activity ：Manual muscle test-8 | About 2 years after LUCAR-DKS1 infusion (Day 1)
  Change in manual muscle testing (MMT-8) score from baseline up to 2 years in IIM patients. This tool assesses muscle strength by testing 8 proximal, distal, and axial muscles ,assess unilateral(score range 0-80 points)handedness side, with a lower score representing a more significant degree of muscle involvement.
SjS disease activity: Sjögren's Tool for Assessing(STAR) | About 2 years after LUCAR-DKS1 infusion (Day 1)
  Proportion and duration of Sjögren's syndrome(r/r SjS) subjects achieving Sjögren's Tool for Assessing Response(STAR) response from baseline up to 2 years. STAR can be used to assess the treatment response of all SjS patients. It is generally believed that a STAR score of ≥ 5 is an effective response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wenfeng Tan Principal Investigator, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (5):
- China (5):
  - The Third The People's Hospital of BengBu, Bengbu, Anhui
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No